CLINICAL TRIAL: NCT07209345
Title: Pre-emptive Scalp Infiltration With Low-dose Flurbiprofen and Ropivacaine for Postoperative Analgesia After Craniotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY-2018-034-02-11
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Post-craniotomy; Pain
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine group (Active Comparator): 0.5% ropivacaine was injected along the planned surgical incision and pin fixation sites of the Mayfield head holder at about 30 min before surgical incision
  Interventions: Drug: Ropivacaine
- FA+Ropivacaine group (Experimental): 5mg FA and 0.5% ropivacaine was injected along the planned surgical incision and pin fixation sites of the Mayfield head holder at about 30 min before surgical incision
  Interventions: Drug: FA+Ropivacaine

INTERVENTIONS:
Drug: FA+Ropivacaine — 0.5 mL FA (50 mg; 5 mL; by Beijing Taide Pharmaceutical Co., Ltd) and 15 mL of 1% ropivacaine (Nai Le Pin 10mg/mL; by AstraZeneca AB, Sweden) diluted to a total volume of 30 mL in normal saline
  Arms: FA+Ropivacaine group
Drug: Ropivacaine — 15 mL of 1% ropivacaine diluted to a total volume of 30 mL in normal saline
  Arms: Ropivacaine group

SUMMARY:
Post-craniotomy pain is common and often associated with poor outcomes. Flurbiprofen axetil (FA) is an injectable NSAID for postoperative analgesia, however, the impact of local FA, remains elusive on post-craniotomy pain. As FA is highly lipophilic by merging into emulsified lipid microspheres, it has a high affinity to the surgical incision and inflammatory tissues to achieve targeted drug therapy and prolonged duration of action. On base of the previous report that local NSAIDs achieved therapeutic tissue concentrations despite a plasma concentration of <5% of that of systemic administration, a low-dose of FA might be considered a preferential option for local infiltration to avoid anti-platelet related side effects, such as intra-cerebral bleeding. In this study, the investigators attempt to evaluate the clinical effects of pre-emptive scalp infiltration with low-dose FA and ropivacaine for postoperative analgesia after craniotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-64 years;
2. ASA physical status of I - II;
3. Scheduled for craniotomy under general anesthesia;
4. Anticipated tracheal extubation, recovery of consciousness and orientation within 2 hours after craniotomy.

Exclusion Criteria:

1. Glasgow Coma Scale <15;
2. Unable to use the PCIA device or comprehend the pain NRS;
3. History of opioid dependence, chronic headache or intake of any drugs with known analgesic properties within the 24 hours before surgery;
4. Any contraindication to flurbiprofen axetil, such as gastrointestinal ulcer, coagulation disorders, renal dysfunction, heart failure and ischemic heart disease;
5. History of allergy to any drug used in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
The cumulative sufentanil consumption (μg) in PCIA device within 48 hours after craniotomy. | within 48 hours after craniotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China